CLINICAL TRIAL: NCT04012567
Title: A Prospective, Multi-center, Randomized Clinical Study to Evaluate the Safety and Effectiveness of Biosure Regenesorb Interference Screw in Arthroscopic Reconstruction of Cruciate Ligaments in Chinese Patients
Brief Title: Safety and Effectiveness of BIOSURE RG in Cruciate Ligaments Reconstruction in Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOSURE RG.SMD.PMA.2019.01
Record Dates: First submitted 2019-06-12; First posted 2019-07-09 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-08

CONDITIONS: Cruciate Ligament Reconstruction; Knee
Keywords: Biosure Regenesorb; Chinese; Cruciate ligaments reconstruction; Prospective; Randomize; Evaluator-blinded

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The Biosure Regenesorb Interference Screw (Experimental): The Biosure Regenesorb Interference Screw, an absorbable screw designed with an open structure and made of biocomposite material, is used to fix ligaments, tendons, soft tissues or bone-tendon-bone grafts in knee surgery.
  Interventions: Device: Investigational device: Biosure Regenesorb Interference Screw
- The BIOSURE HA Interference Screw (Active Comparator): The Biosure HA Interference Screw, an absorbable screw made of biocomposite material, is used to fix ligaments, tendons, soft tissues or bone-tendon-bone grafts in knee surgery.
  Interventions: Device: Control device: BIOSURE HA Interference Screw

INTERVENTIONS:
Device: Investigational device: Biosure Regenesorb Interference Screw — The Biosure Regenesorb Interference Screw, an absorbable screw designed with an open structure and made of biocomposite material made of PLGA, β-TCP and calcium sulfate, is used to fix ligaments, tendons, soft tissues or bone-tendon-bone grafts in knee surgery. Its open structural design enables rapid bone ingrowth to make the screw integrated with bone tissues so as to promote healing.
  Arms: The Biosure Regenesorb Interference Screw
Device: Control device: BIOSURE HA Interference Screw — BIOSURE HA Interference Screws and Drivers are designed for durability and reduced screw breakage. Both the screws and driver have been enhanced to allow screws to fully seat on the driver all the way to the tip of the screw, helping stress distribution and force transfer. The screw design also incorporates a consistent wall thickness throughout the length of the screw for added durability and features a tapered body for ideal ease of insertion.
  Arms: The BIOSURE HA Interference Screw

SUMMARY:
The objective of this study is to compare the safety and effectiveness of Biosure Regenesorb Interference Screw versus BIOSURE HA Interference Screw (control device) in patients requiring reconstruction of cruciate ligaments of the knee. The trial results will be used for registration of Biosure Regenesorb Interference Screw in China.

The primary efficacy endpoint of this study is Lysholm score at 12 months after operation. The non-inferiority testing is performed for efficiency of primary efficacy endpoint, and the test hypothesis is as follows:

Invalid hypothesis: H0: μ1-μ2 ≤-δ Alternative hypothesis: H1: μ1-μ2 > -δ, where, μ1 and μ2 are the Lysholm scores in the investigational group and control group, respectively. δ is a non-inferiority critical value.

DETAILED DESCRIPTION:
The clinical trial is designed to be a prospective, multi-center, randomized, evaluator-blinded, parallel-controlled, non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the inclusion criteria:

  1. Signing the Informed Consent Form (ICF) voluntarily;
  2. Patients aged 18-75 years;
  3. Patients clinically diagnosed with knee cruciate ligaments rupture or tear and suitable for cruciate ligaments reconstruction definitely;
  4. Normal contralateral knee joint.

Exclusion Criteria:

* Subjects with any of the following characteristics must be excluded from participation in the study:

  1. Patients not complying with the diagnosis criteria for cruciate ligaments rupture or tear;
  2. Patients with an unclosed epiphyseal plate shown on the X-ray film;
  3. Patients having underwent internal fixation or reconstruction due to a knee joint fracture;
  4. Patients with obvious knee joint degeneration shown on the X-ray film;
  5. Patients who cannot make a knee flexion of not less than 90° during operation;
  6. Patients undergoing autologous chondrocyte implantation;
  7. Patients with medial meniscus or lateral meniscus completely resected;
  8. Patients with significant anatomical abnormalities;
  9. Pregnant or breast-feeding females or those at a child-bearing age planning to become pregnant;
  10. Patients with serious osteoporosis that affects screw implantation;
  11. Patients with a malignant tumor that causes failure to effectively fix the implant;
  12. Known hypersensitivity to the implant materials;
  13. Patients not suitable for operation due to obvious local or systemic infection;
  14. Patients who cannot tolerate an operation due to severe malnutrition;
  15. Patients with severe coagulation disorder (judged by the investigator), e.g. the hemophiliac;
  16. Patients with immunodeficiency, including those who must receive immunosuppressant for a long time;
  17. Patients with extensive skin diseases;
  18. Obese patients having a Body Mass Index (BMI) > 35;
  19. Patients who cannot cooperate in postoperative rehabilitation due to a severe mental disease or those who cannot tolerate the operation due to a cardiopulmonary disease;
  20. Patients who received operation on the injured lower limb within the past 1 year;
  21. Patients who participated in any other clinical trial within the past three months;
  22. Patients who cannot follow the requirements described in the study protocol; and
  23. Other patients who are considered by the investigator not suitable for this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi Gong, Professor, Principal Investigator — Peking University Third Hospital
Locations (4):
- China (4):
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Third Hospital, Beijing, Haidian District
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant enrolled in the study was excluded because their cruciate ligament was found to be unbroken during operation.
Period: Overall Study
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Started | 69 | 70
Completed | 68 | 69
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.12 (8.90) | 33.69 (9.89) | 31.91 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 54 | 57 | 111
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.31 (3.29) | 24.78 (3.14) | 24.55 (3.21)

OUTCOME MEASURES:

1. Primary Outcome: Lysholm Knee Scoring Scale 12 Months After Operation
Description: Lysholm Knee Scoring Scale evaluates functions of participants based on 8 items: limp, support, interlocking, pain, instability, swelling, stair climbing and squatting. The total Lysholm score is 0-100. Pain and instability account for a higher proportion in this score. The knee functions of patients are considered excellent when the score is 95-100, good when 84-94, fair when 65-83 and poor when less than 65 (i.e., 100 is best outcome and 0 is the worst outcome).
Time Frame: 12 months
Population: Full Analysis Set (FAS) included participants with at least one effectiveness evaluation that provided data for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 69 | 70
score on a scale | 92.49 (10.61) | 94.14 (7.13)

2. Secondary Outcome: Lysholm Knee Scoring Scale Pre-Operation and 6 Months & 24 Months After Operation
Description: as for outcome 1
Time Frame: Pre-Operation, Post-Operation 6 months, 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 69 | 70
score on a scale
  Pre-Operation | 72.42 (14.41) | 70.19 (16.61)
  Post-Operation 6 months: number analyzed (Participants) | 69 | 69
  Post-Operation 6 months | 87.35 (12.54) | 87.14 (11.67)
  24 months: number analyzed (Participants) | 68 | 69
  24 months | 94.22 (8.46) | 94.96 (7.32)

3. Secondary Outcome: International Knee Documentation Committee (IKDC) Score
Description: The International Knee Documentation Committee (IKDC) score is composed of a knee evaluation form (10 items) and a knee ligament examination form (8 items), involving joint pain, sport level and ability of daily activities. The total score is transformed to a scale ranging from 0 to 100, where 0 represents the lowest level of knee function and highest level of symptoms (i.e., worst outcome), and 100 represents the highest level of knee function and lowest level of symptoms (i.e., best outcome).
Time Frame: Pre-Operation, Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 69 | 70
score on a scale
  Pre-Operation | 66.75 (12.95) | 65.50 (15.41)
  Post-Operation 6 months: number analyzed (Participants) | 69 | 69
  Post-Operation 6 months | 80.98 (8.07) | 80.01 (8.60)
  12 months: number analyzed (Participants) | 68 | 69
  12 months | 88.83 (9.24) | 91.00 (7.45)
  24 months: number analyzed (Participants) | 68 | 69
  24 months | 91.41 (8.38) | 92.90 (6.87)

4. Secondary Outcome: Drawer Test: Anterior
Description: The Anterior Drawer Test is used for anterior cruciate ligament (ACL) examination with an outcome of either negative or positive. The test was performed with the participant lying supine with the knee flexed at 90 degrees and the foot stabilized flat on the table. The examiner then grasped the tibia and applied an anterior force to assess displacement. The test outcome was measured by the number of participants with a negative or positive result. A positive test indicated forward straight instability, defined as the tibia being displaced forward by 5 millimeters (mm) or more compared to the uninjured side.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 68 | 67
Participants
  Post-Operation 6 months: Negative | 68 | 67
  Post-Operation 6 months: Postive | 0 | 0
  12 months: number analyzed (Participants) | 61 | 67
  12 months: Negative | 61 | 67
  12 months: Postive | 0 | 0
  24 months: number analyzed (Participants) | 53 | 61
  24 months: Negative | 53 | 61
  24 months: Postive | 0 | 0

5. Secondary Outcome: Drawer Test: Posterior
Description: The Posterior Drawer Test is used for posterior cruciate ligament (PCL) examination with an outcome of either negative or positive. The test was performed with the participant lying supine with the knee flexed at 90 degrees. The examiner placed both hands on the proximal lower leg (just below the knee joint) with thumbs on the tibial tuberosity then attempted to translate the lower leg posteriorly. The test outcome was measured by the number of participants with a negative or positive result. A positive test indicated a lack of end feel or excessive posterior translation.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 68 | 67
Participants
  Post-Operation 6 months: Negative | 68 | 66
  Post-Operation 6 months: Positive | 0 | 1
  12 months: number analyzed (Participants) | 61 | 67
  12 months: Negative | 61 | 67
  12 months: Positive | 0 | 0
  24 months: number analyzed (Participants) | 49 | 57
  24 months: Negative | 49 | 57
  24 months: Positive | 0 | 0

6. Secondary Outcome: Lachman Test
Description: The Lachman Test assessed integrity of the anterior cruciate ligament (ACL) with an outcome of either negative or positive. The test was performed with the participant lying supine with the knee flexed to 20-30 degrees and the injured limb slightly rotated outward. The examiner immobilized the lower end of the femur with one hand and pressed the posterior side of the upper end of the tibia forward or backward. The test outcome was measured by the number of participants with a negative or positive result. A positive test indicated excessive anterior translation of the tibia greater than the uninjured side along with a soft end feel.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 68 | 67
Participants
  Post-Operation 6 months: Negative | 68 | 67
  Post-Operation 6 months: Positive | 0 | 0
  12 months: number analyzed (Participants) | 61 | 67
  12 months: Negative | 61 | 67
  12 months: Positive | 0 | 0
  24 months: number analyzed (Participants) | 53 | 61
  24 months: Negative | 53 | 61
  24 months: Positive | 0 | 0

7. Secondary Outcome: Imaging Evaluation: X-ray
Description: Radiographic assessment taken from x-ray images to evaluate the general view of bone. The assessment measured the number of participants categorized with either a normal or abnormal imaging evaluation.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 67 | 66
Participants
  Post-Operation 6 months: Normal | 0 | 1
  Post-Operation 6 months: Abnormal | 67 | 65
  12 months: number analyzed (Participants) | 61 | 65
  12 months: Normal | 1 | 1
  12 months: Abnormal | 60 | 64
  24 months: number analyzed (Participants) | 51 | 61
  24 months: Normal | 0 | 0
  24 months: Abnormal | 51 | 61

8. Secondary Outcome: Imaging Evaluation: Computed Tomography (CT)
Description: Radiographic assessment taken from Computed Tomography (CT) images to evaluate specific view of bone. The assessment measured the number of participants categorized with either a normal or abnormal imaging evaluation.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 67 | 66
Participants
  Post-op 6 months: Normal | 0 | 0
  Post-op 6 months: Abnormal | 67 | 66
  12 months: number analyzed (Participants) | 61 | 66
  12 months: Normal | 0 | 0
  12 months: Abnormal | 61 | 66
  24 months: number analyzed (Participants) | 50 | 61
  24 months: Normal | 0 | 0
  24 months: Abnormal | 50 | 61

9. Secondary Outcome: Imaging Evaluation: Magnetic Resonance Imaging (MRI)
Description: Radiographic assessment taken from Magnetic Resonance Imaging (MRI) to evaluate ligament. The assessment measured the number of participants categorized with either a normal or abnormal imaging evaluation.
Time Frame: Post-Operation 6 months, 12 months, 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
Number analyzed (Participants) | 68 | 67
Participants
  Post-Operation 6 months: Normal | 0 | 0
  Post-Operation 6 months: Abnormal | 68 | 67
  12 months: number analyzed (Participants) | 61 | 67
  12 months: Normal | 0 | 0
  12 months: Abnormal | 61 | 67
  24 months: number analyzed (Participants) | 52 | 62
  24 months: Normal | 0 | 0
  24 months: Abnormal | 52 | 62

ADVERSE EVENTS:
Time Frame: Adverse events were collected upon device implantation through 24 months, approximately 740 days.
Arm/Group | The Biosure Regenesorb Interference Screw | The BIOSURE HA Interference Screw
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/69 | 3/70
Other Adverse Events (participants affected / at risk) | 30/69 | 26/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | The Biosure Regenesorb Interference Screw (N=69) | The BIOSURE HA Interference Screw (N=70)
Prepuce balanitis, prepuce too long (General disorders) | 1 | 0 — definitely not related to device
Meniscus Injury of the right knee (Injury, poisoning and procedural complications) | 0 | 1 — possibly related to the device
Left knee anterior cruciate ligament rupture,lateral meniscus root tear (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
Foreign body reaction (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
Thrombosis:middle & lower left superficial femoral, popliteal, posterior tibial,& intermuscular vein (Vascular disorders) | 1 | 0 — definitely not related to device
Pharyngeal disorder (General disorders) | 0 | 1 — definitely not related to device
Anterior cruciate ligament injury in right knee, meniscus injury in right knee (Musculoskeletal and connective tissue disorders) | 0 | 1 — definitely not related to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | The Biosure Regenesorb Interference Screw (N=69) | The BIOSURE HA Interference Screw (N=70)
INJURY OF POSTERIOR HORN OF MENISCUS ON THE LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
WOUND PAIN (General disorders) | 4 | 0 — possibly related to the device
FLAT WART (Skin and subcutaneous tissue disorders) | 1 | 0 — definitely not related to device
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
ALLERGY (Immune system disorders) | 0 | 1 — possibly related to the device
PERIFOLLICULAR KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 1 — definitely not related to device
WOUND PAIN (General disorders) | 0 | 6 — possibly related to the device
HYPERCHOLESTEROLEMIA (Endocrine disorders) | 0 | 1 — definitely not related to device
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
SYMPTOMS OF LOW GRADE FEVER (General disorders) | 1 | 0 — definitely not related to device
HYPERURICEMIA (Renal and urinary disorders) | 1 | 0 — possibly related to the device
ACROMIAL IMPINGEMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 — definitely not related to device
SWELLING OF LEFT KNEE (General disorders) | 0 | 1 — possibly related to the device
RIGHT PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
UPPER RESPIRATORY INFECTION (URI) (Infections and infestations) | 0 | 1 — definitely not related to device
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0 — possibly related to the device
LIGAMENT STRAIN IN LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
INSOMNIA (Nervous system disorders) | 1 | 0 — definitely not related to device
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 1 | 0 — definitely not related to device
LEFT PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
POSTOPERATIVE ANESTHESIA GASTROINTESTINAL REACTION (Gastrointestinal disorders) | 1 | 0 — definitely not related to device
POSSIBLE HYPOGLYCAEMIA (Endocrine disorders) | 1 | 0 — possibly related to the device
FEVER (General disorders) | 0 | 1 — possibly related to the device
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — definitely not related to device
FREQUENT URINATION (Renal and urinary disorders) | 1 | 0 — definitely not related to device
QUADRICEPS ATROPHY (Musculoskeletal and connective tissue disorders) | 0 | 3 — possibly related to the device
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
LARYNGOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — definitely not related to device
ANXIETY STATE (Psychiatric disorders) | 1 | 0 — definitely not related to device
SOFT TISSUE STRAINS OF RIGHT FOOT (General disorders) | 1 | 0 — definitely not related to device
SWELLING IN THE LEFT KNEE (General disorders) | 1 | 0 — possibly related to the device
QUADRICEPS ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
INFLAMMATION (General disorders) | 0 | 1 — definitely not related to device
RIGHT KNEE OSTEOARTHRITIS AGGRAVATED (Musculoskeletal and connective tissue disorders) | 0 | 1 — definitely not related to device
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 | 2 — definitely not related to device
CONJUNCTIVITIS OF THE RIGHT EYE (Eye disorders) | 0 | 1 — definitely not related to device
NASAL BLEEDING (Vascular disorders) | 0 | 1 — definitely not related to device
INCISION REDNESS AND SWELLING (Skin and subcutaneous tissue disorders) | 0 | 1 — possibly related to the device
HEADACHE (Nervous system disorders) | 0 | 1 — definitely not related to device
DIZZINESS (Nervous system disorders) | 0 | 1 — definitely not related to device
SYNOVITIS OF THE RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
FOCAL NODULAR HYPERPLASIA OF LIVER (Hepatobiliary disorders) | 0 | 1 — definitely not related to device
DISUSE OSTEOPOROSIS OF THE RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 0 | 2 — possibly related to the device
RIGHT QUADRICEPS FEMORIS MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
SWELLING IN THE RIGHT KNEE (General disorders) | 0 | 1 — possibly related to the device
LEFT QUADRICEPS ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
SLIGHT SWELLING OF THE LEFT KNEE JOINT (General disorders) | 1 | 0 — possibly related to the device
SYMPTOMS OF FEVER (General disorders) | 1 | 0 — possibly related to the device
SOFT TISSUE CONTUSION OF LEFT KNEE (Injury, poisoning and procedural complications) | 1 | 0 — possibly related to the device
TENOSYNOVITIS STENOSANS OF STYLOID PROCESS OF RADIUS OF LEFT WRIST (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
IRREGULAR PERIODS (Reproductive system and breast disorders) | 1 | 0 — definitely not related to device
FALL INDUCED PAIN IN RIGHT KNEE JOINT FOR 3 DAYS (Injury, poisoning and procedural complications) | 1 | 0 — definitely not related to device
NUMBNESS IN THE MEDIAL LEG (Nervous system disorders) | 1 | 0 — definitely not related to device
ANTERIOR TISSUE SWELLING OF RIGHT KNEE (General disorders) | 1 | 0 — definitely not related to device
PAIN IN THE RIGHT KNEE JOINT CAUSED BY SPRAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
BONE MARROW TUNNEL CYST OF THE RIGHT KNEE TIBIA (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
FEVER SYMPTOM (General disorders) | 0 | 1 — definitely not related to device
ECZEMATOID DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 — possibly related to the device
CHRONIC PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — definitely not related to device
POSTOPERATIVE DYSFUNCTION OF LEFT KNEE JOINT TRAUMA (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
PAIN IN THE WOUND (General disorders) | 1 | 0 — possibly related to the device
ATROPHY OF THE QUADRICEPS FEMORIS OF THE LEFT LOWER EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 — possibly related to the device
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 1 | 0 — definitely not related to device
TRAUMATIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
FOREIGN BODY REACTION (General disorders) | 1 | 0 — possibly related to the device
INFLAMMATION (Musculoskeletal and connective tissue disorders) | 0 | 1 — definitely not related to device
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 — definitely not related to device
THROMBOSIS OF RIGHT LOWER EXTREMITY (Vascular disorders) | 1 | 0 — possibly related to the device
PALPITATE (Cardiac disorders) | 0 | 1 — definitely not related to device
HYPERLIPIDEMIA WITH ATHEROSCLEROSIS (Vascular disorders) | 0 | 1 — definitely not related to device
HYPERTENSION (General disorders) | 0 | 1 — definitely not related to device
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 0 — definitely not related to device
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 — definitely not related to device
SWELLING OF SOFT TISSUE AROUND THE LEFT KNEE (General disorders) | 1 | 0 — definitely not related to device
SCROTAL INFLAMMATION (Skin and subcutaneous tissue disorders) | 1 | 0 — definitely not related to device
LEFT KNEE CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 — definitely not related to device
DISUSE OSTEOPOROSIS OF THE LEFT KNEE (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
RIGHT KNEE PAIN (General disorders) | 0 | 1 — definitely not related to device
RIGHT KNEE EFFUSION (General disorders) | 0 | 1 — possibly related to the device
SWELLING IN THE RIGHT LOWER EXTREMITY (General disorders) | 0 | 2 — possibly related to the device
OOR MOTION OF THE RIGHT KNEE JOINT (LACK OF EXERCISE AFTER SURGERY) (Musculoskeletal and connective tissue disorders) | 0 | 1 — possibly related to the device
QUADRICEPS ATROPHY OF THE RIGHT LOWER LIMB (Injury, poisoning and procedural complications) | 0 | 1 — possibly related to the device
RIGHT RADIAL STYLOIDITIS (General disorders) | 0 | 1 — definitely not related to device
CHRONIC VAGINITIS (Infections and infestations) | 0 | 1 — definitely not related to device
SKIN PAPILLOMA（ FLAT WARTS) (Skin and subcutaneous tissue disorders) | 1 | 0 — definitely not related to device
POSTOPERATIVE JOINT HEMATOMA (Vascular disorders) | 0 | 1 — definitely not related to device
CHRONIC PROSTATITIS (General disorders) | 1 | 0 — definitely not related to device
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 1 | 0 — definitely not related to device
THYROID NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — definitely not related to device
SECONDARY OLIGOMENORRHEA (Reproductive system and breast disorders) | 1 | 0 — definitely not related to device
FEVER (General disorders) | 1 | 0 — possibly related to the device
ANTERIOR TISSUE SWELLING OF RIGHT KNEE (General disorders) | 0 | 1 — definitely not related to device
KNEE PAIN IN RIGHT KNEE (General disorders) | 0 | 1 — definitely not related to device
MAMMARY PAIN (General disorders) | 1 | 0 — definitely not related to device
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 — definitely not related to device
RIGHT QUADRICEPS ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0 — definitely not related to device
ACUTE UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 — definitely not related to device
CAT SCRATCH (Injury, poisoning and procedural complications) | 0 | 1 — definitely not related to device
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 1 — definitely not related to device
URINE OCCULT BLOOD (Renal and urinary disorders) | 0 | 1 — definitely not related to device
VERRUCA VULGARIS (Skin and subcutaneous tissue disorders) | 0 | 1 — definitely not related to device
ABDOMINAL PAIN (General disorders) | 0 | 1 — definitely not related to device
CONJUNCTIVITIS OF BOTH EYES (Eye disorders) | 0 | 1 — definitely not related to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT04012567/Prot_SAP_000.pdf